CLINICAL TRIAL: NCT03357861
Title: Characteristics and Care of Solid Tumor Patients Treated With Immunotherapy Admitted in Intensive Care Unit.
Brief Title: Cancer Patients Treated With Immunotherapy in Intensive Care Unit
Acronym: IMMUNO-REA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.290
Record Dates: First submitted 2017-11-17; First posted 2017-11-30 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Cancer; Critical Illness; Immunotherapy
Keywords: cancer; intensive care unit; checkpoint inhibitors; adverse event
MeSH Terms: conditions — Neoplasms; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This work aims to describe the characteristics and methods of management of patients suffering from a solid tumor treated with immunotherapy admitted to intensive care.

DETAILED DESCRIPTION:
The place of checkpoint inhibitors (anti-PD-1 and PD-L-1) is currently validated in the management of melanoma and metastatic non-small cell lung cancer. The toxicity profile is specific with adverse effects related to immunity. Some side effects (myocarditis, colitis, interstitial lung disease, etc.) can be severe and patient could be hospitalized in intensive care unit.

The question of immunotherapy's imputability in the acute disease is becoming more frequent.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years old;
* with a solid tumor;
* Treatment with anti-CTLA4 and / or anti-PD-1 / PDL-1 still in progress or up to 6 months after stopping;
* Admitted to resuscitation or continuous care in an unprogrammed way, whatever the reason.

Exclusion Criteria:

* Minors;
* Pregnant or lactating woman;
* Admission after surgery of a scheduled surgery or for the security of procedure;
* Anti-CTLA4 and / or anti-PD-1 / PDL-1 treatment stopped for more than 6 months;
* Subject under guardianship or deprivation of liberty;
* Refusal of consent;
* No affiliation to a health insurance scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated with anti-CTLA4 and/or anti-PD-1 / anti-PD-L1 or up to 6 months after stopping admitted in ICU
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the imputability of immunotherapy in the ICU admission reason for lung cancer patients treated by immunotherapy. | At ICU discharge (maximum 30 days)
  Description of ICU admission reason (immunotherapy toxicity versus other) for lung cancer patients treated by immunotherapy

SECONDARY OUTCOMES:
Description of the immunosuppressive treatments prescribed during the stay in intensive care for the patient's care. | At ICU discharge (maximum 30 days)
  immunosuppressive treatments in intensive care unit
Description of ICU survival | At ICU discharge (maximum 60 days)
  ICU survival
Description of hospital survival | At hospital discharge (maximum 60 days)
  Hospital survival

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire TOFFART, MD-PhD, Principal Investigator — UniversityHospital Grenoble
Locations (2):
- Institut Jules Bordet, Brussels, Belgium
- UniversityHospitalGrenoble, Grenoble, France